CLINICAL TRIAL: NCT03763604
Title: Named Patient Use Program to Provide Abemaciclib for the Treatment of Metastatic Breast Cancer
Brief Title: Named Patient Use Program to Provide Abemaciclib (LY2835219) for the Treatment of Metastatic Breast Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 17088; I3Y-MC-Y001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Abemaciclib — Administered orally.
  Other Names: LY2835219

SUMMARY:
The treating physician/investigator contacts Lilly when, based on their medical opinion, a patient meets the criteria for inclusion in the expanded access program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hormone receptor positive metastatic breast cancer for whom there is reasonable expectation that abemaciclib may provide clinical benefit and who are suitable to receive abemaciclib.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (160):
- Australia (20):
  - Liverpool Hospital, Liverpool, New South Wales
  - North West Cancer Centre, North Tamworth, New South Wales
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Mater Hospital Sydney, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Adelaide Oncology and Haematology, Calvary Central Districts Hospital, Elizabeth Vale, South Australia
  - Icon Cancer Centre - Hobart, Hobart, Tasmania
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital Outpatients, Box Hill, Victoria
  - Epworth Eastern Hospital, Box Hill, Victoria
  - Melbourne Cancer Care, Brighton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Dr. Zimet Private Room, Richmond, Victoria
  - Slade Pharmacy Epworth Hospital, Richmond, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Icon Cancer Care - The Wesley Medical Centre, Auchenflower
  - Northern Beaches Hospital, Freches Forest
  - South Coast District Hospital, Victor Harbor
- Canada (11):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Vancouver, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island, Victoria, British Columbia
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Unity Health Toronto, St. Michael's Hospital, Toronto, Ontario
  - CHUL du CHU de Québec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Cairo Oncology Center (Cairo Cure), Mohandeseen, Cairo Governorate, Egypt
- India (2):
  - Apollo Cancer Institute, Apollo Speciality Hospital, Teynampet, Chennai
  - Indraprastha Apollo Hospital, New Delhi
- Italy (3):
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Torre, Roma
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
  - Ospedale Di Circolo E Fondazione Macchi, Varese
- Malaysia (14):
  - Pantai Hospital Sungai Petani, Sungai Petani, Kedah
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - Beacon Hospital, Off Jalan Templer, Petaling JAYA
  - Pantai Hospital Penang, Bayan BARU, Pulau Pinang
  - Gleneagles Penang, George Town, Pulau Pinang
  - Loh Guan Lye Specialists' Centre, George Town, Pulau Pinang
  - Penang Adventist Hospital, George Town, Pulau Pinang
  - Mount Miriam Cancer Hospital, Tanjung Bungah, Pulau Pinang
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Subang Jaya Medical Centre, Petaling Jaya, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Universiti Malaya Medical Centre, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Institut Kanser Negara, Putrajaya
- Elizabeth Au Oncology, Singapore, Singapore
- South Africa (15):
  - Vincent Pallotti Hospital, Pinelands, Cape Town
  - Flora Clinic, Floracliff, Gauteng
  - Olivedale Clinic, Johannesburg, Gauteng
  - Netcare Linksfield Hospital, Johannesburg, Gauteng
  - Donald Gordon Medical Center, Johannesburg, Gauteng
  - Wits Donald Gordon Clinical Trial Center, Johannesburg, Gauteng
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Sandton Oncology, Morningside, Gauteng
  - DGMC Oncology, Parktown, Gauteng
  - Amanzimtoti Oncology Centre, Durban, KwaZulu-Natal
  - Hopelands Cancer Centre Hilton, Hilton, KwaZulu-Natal
  - Abraham Oncology, Richards Bay, KwaZulu-Natal
  - Cancercare, George, Western Cape
  - Cancercare Rondebosch Oncology, Cape Town
  - Dr Pirjol and Szpak Inc. Oncology Pratice, eManzimtoti
- South Korea (17):
  - National Cancer Center, Ilsandong-gu, Goyang-si Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Inha University Hospital, Incheon, Incheon-gwangyeoksi [Incheon]
  - St. Mary's Hospital, Gyeonggi-do, Korea
  - Gachon University Gil Medical Center, Namdong-gu, Incheon, Korea
  - Seoul St. Mary's Hospital, Seoul, Korea
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul, Korea
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Ewha University Mokdong Hospital, Seoul, Yangcheon-gu
  - Chungbuk National University Hospital, Chungcheongbuk-do
  - Kyungpook National University Medical Center Chilgok Hospital, Daegu
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (42):
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona [Barcelona]
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona, Barcelona
  - Institut Catala d'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Duran I Reynals, L'Hospitalet de Llobregat, Barcelona
  - Corporacion Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Germans Trias i Pujol, Badalona, Catalunya [Cataluña]
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, La Laguna
  - Hospital la Zarzuela, Aravaca, Madrid
  - Hospital De Mostoles, Móstoles, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Son Espases, Palma de Mallorca, Palma de Mallorca(Baleares)
  - H. San Francisco de Borja (H. GANDIA), Gandia, Valencia
  - Hospital Lluis Alcanyis, Xàtiva, Valencia
  - Hospital De Basurto, Bilbao, Vizcaya
  - Hospital Arquitecto Marcide (Área Sanitaria de Ferrol), A Coruña
  - Hospital General de Albacete, Albacete
  - Hospital Quironsalud Barcelona- END, Barcelona
  - Hospital Quirón Salud Barcelona-Instituto Oncológico Baselga, Barcelona
  - Hospital Universitari Dexeusa, Barcelona
  - Instituto Oncologico Dr Rosell (IOR), Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario San Cecilio, Granada
  - Cl. Universitaria Navarra, Madrid
  - Centro Oncológico MD Anderson, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Hospital Infanta Cristina, Madrid
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Clinico Universitario Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova Valencia, Valencia
  - Hospital Doctor Peset, Valencia
  - Hospital de Sagunto, Valencia
  - IDCQ HOSPITALES Y SANIDAD, S.L.U. (Hospital Quirón Zaragoza), Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
  - Hospital Universitario Zaragoza, Zaragoza
- Switzerland (10):
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Hôpital de la Tour, La Tour Hôpital Privé SA, Meyrin, Canton of Geneva
  - Tumorzentrum ZeTuP Rapperswil-Jona, Rapperswil, Canton of St. Gallen
  - Tumor- und Brustzentrum ZeTuP Sankt Gallen, Sankt Gallen, Canton of St. Gallen
  - Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - Oncologia Varini Calderoni Christinat, Lugano, Canton Ticino
  - Hôpitaux Universitaires de Genève, Geneva
  - HUG-Hôpitaux Universitaires de Genève, Geneva
  - Luzerner Kantonsspital, Lucerne
  - OnkoZentrum Zürich AG, Zurich
- Taiwan (16):
  - Chiayi Chang Gung Memorial Hospital, Putzu City, Chiayi County
  - Kaohsiung Chang Gung Memorial Hospital, Niaosong Dist, Kaohsiung City
  - Tri-Service General Hospital, Taipei City, Taipei
  - National Taiwan University Hospital Yunlin Branch, Zhongzheng District, Taipei
  - MacKay Memorial Hospital, New Taipei City, Tamsui District
  - Taichung Tzu Chi Hospital, Taichung, Tanzi District
  - Saint Paul's Hospital, Taoyuan District, Taoyuan District
  - National Taiwan University Hospital Yunlin Branch, Yunlin County, Douliu City, Yunlin County, Douliu City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Municipal Siaogang Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yan-Sen Cancer Center, Taipei
- Thailand (5):
  - Songklanagarind Hospital, Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital, Muang Chiangmai, Chiangmai
  - Rajavithi Hospital, Bangkok, Ratchathewi District
  - King Chulalongkorn Memoiral Hospsital, Bangkok
  - Ramathibodi Hopsital, Bangkok
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Loom Dene, Radlett, Hertfordshire
  - Northern Centre for Cancer Treatment, Newcastle upon Tyne, Tyne and Wear